CLINICAL TRIAL: NCT03526731
Title: Quadratus Lumborum Block for Postoperative Pain Control in Patients Undergoing Unilateral Inguinal Hernia Repair, a Comparative Study Between Two Approaches
Brief Title: Analgesic Efficacy of Trans-muscular Quadratus Lumborum Block After Unilateral Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia and SICU - Faculty of Medicine - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-13-2016
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain; Ultrasound Guided Nerve Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (original QLB-2): (Experimental): Local anesthetic will be injected between the quadratus lumborum muscle and the latissimus dorsi muscle guided by ultrasound.
  Interventions: Other: ultrasound guided quadratus lumborum block
- Group B (trans-muscular OLB-3) (Experimental): Local anesthetic will be injected between quadratus lumborum and psoas major after passing through the quadratus lumborum muscle guided by ultrasound.
  Interventions: Other: ultrasound guided quadratus lumborum block

INTERVENTIONS:
Other: ultrasound guided quadratus lumborum block — ultrasound guided quadratus lumborum block for post operative pain control after unilateral inguinal hernia repair.

SUMMARY:
A significant component of pain experienced after abdominal surgery is related to incision of the abdominal wall and adequate analgesia can be a challenge.

The ultrasound-guided (USG) quadratus lumborum block QLB was first described by Rafael Blanco in a presentation at ESRA 2007 at the XXVI Annual ESRA Congress in Valencia, Spain. Blanco described a potential space posterior to the abdominal wall muscles and lateral to the quadratus lumborum muscle where Local anesthetics can be injected. This technique provide analgesia after abdominal surgery due to spread of LA from its lumbar deposition cranially into the thoracic paravertebral space where lateral and anterior cutaneous branches from Th7 to L1 can be blocked . This was proved by Carney et al. who found traces of contrast agent in the TPVS following application of this block A novel USG QL block is the transmuscular approach which relies on clearly identifiable sonographic bony landmarks, Where the needle is advanced through the QL muscle, penetrating the ventral proper fascia of the QL muscle and LA is finally injected between the QL and Psoas major (PM) muscle. The transmuscular QL block does not result in redundant antero-lateral spread of the injectate. This may indicate that lower volumes of LA potentially can be used and yet provide extensive thoracolumbar anesthesia.

This study was designed to compare the duration of analgesia provided by the original QLB and transmuscular QLB in patients undergoing surgical repair of unilateral inguinal hernia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II, scheduled for unilateral inguinal hernia repair

Exclusion Criteria:

* Patients with systemic hypertension, cardiovascular disease, cerebrovascular insufficiency, coagulation abnormities, renal or hepatic insufficiency, infection at the injection site, strangulated hernia and hypersensitivity to the local anesthetics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
duration of block | immediately after the end of LA injection till patients pain complaint (VAS > 3) over a period of 24 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Ahmed, MD, Principal Investigator — Faculty of Medicine - Cairo University _ Egypt
Locations (1):
- Abeer Ahmed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Ahmed A, Fawzy M, Nasr MAR, Hussam AM, Fouad E, Aboeldahb H, Saad D, Osman S, Fahmy RS, Farid M, Waheb MM. Ultrasound-guided quadratus lumborum block for postoperative pain control in patients undergoing unilateral inguinal hernia repair, a comparative study between two approaches. BMC Anesthesiol. 2019 Oct 17;19(1):184. doi: 10.1186/s12871-019-0862-z. PMID 31623572